CLINICAL TRIAL: NCT05677841
Title: Investigation of the Effects of Spinal Stabilization Exercises Focusing on the Pelvic Floor in Women With Overactive Bladder
Brief Title: Effects of Spinal Stabilization Exercises Focusing on the Pelvic Floor in Women With Overactive Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, seyda toprak celenay, associate professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/12/23
Record Dates: First submitted 2022-12-29; First posted 2023-01-10 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Exercise group will be given spinal stabilization exercises focusing on the pelvic floor and lifestyle reccommendations
  Interventions: Other: Stabilization exercise+lifestyle recommendation
- Control group (Active Comparator): Control group will be given lifestyle recommendations
  Interventions: Other: lifestyle recommendations

INTERVENTIONS:
Other: Stabilization exercise+lifestyle recommendation — Exercise program was given both spinal stabilization exercises focusing on the pelvic floor 3 days a week for eight weeks and a booklet related to the lower urinary system symptoms, the structure of the pelvic floor and healthy behavioral strategies recommendations (fluid intake, diet, weight control etc. )
  Arms: Exercise group
Other: lifestyle recommendations — The control group will be given a booklet related to the lower urinary system symptoms, the structure of the pelvic floor and healthy behavioral strategies recommendations (fluid intake, diet, weight control etc. )
  Arms: Control group

SUMMARY:
The aim of this study is to examine the effects of spinal stabilization exercises focusing on the pelvic floor on urinary symptoms, spinal stability, pelvic floor muscle functions, quality of life and perception of recovery in women with overactive bladder.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is defined by the International Continence Society and the International Society of Urogynecology as urinary urgency with or without urinary incontinence, usually accompanied by frequency and nocturia. Among the treatment options of OAB; first-line treatments include lifestyle recommendations, exercise approaches, and bladder training. Lifestyle recommendations; healthy lifestyle includes behavioral changes. Spinal stabilization exercise also aims to improve the neuromuscular control, strength and endurance of the muscles that are important in maintaining trunk stability. In recent years, it has been stated that trunk stability is impaired in women with OAB. However, no study was found on spinal stabilization exercises in patients with OAB.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Women with a diagnosis of overactive bladder
* Women who volunteered to participate in the study

Exclusion Criteria:

* Women with only stress urinary incontinence
* Presence of advanced pelvic organ prolapse
* Having a mental problem that will prevent cooperation in assessment and/or practices
* Women with the presence of a malignant condition
* Concomitant neurological disease and/or neurogenic bladder
* Presence of infection
* Pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with overactive bladder
Enrollment: 40 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Overactive bladder symptoms | change from baseline at 8 weeks
  The Overactive Bladder Questionnaire -V8 will be used for the overactive bladder symptoms severity. It has 8 items and the total score can range from 0 to 40. As the score increases, the severity of symptoms increases.

SECONDARY OUTCOMES:
Bladder function | change from baseline at 8 weeks
  Voiding dairy will be used to evaluate the bladder function. In the diary, women will be asked to record some parameters such as voiding time and volume, number of UI, and the amount and type of fluid intake.
Urgency severity | change from baseline at 8 weeks
  Patients' Perception of Intensity of Urgency Scale will be used to evaluate urgency severity.
  According to this scale, "0" means no sense of urgency, "1" means mild urge to urinate, "2" means moderate urge to urinate, "3" means severe urge to urinate, and "4" means urge type incontinence.
Spinal stability | change from baseline at 8 weeks
  The Sharman test will be used to evaluate spinal stability. In this test, the inflatable pad of a pressure biofeedback unit was placed in the natural lordotic curve of the back and was inflated to 40mmHg whilst the subject is lying supine. The subject will be activated the stabilising musculature via the abdominal bracing technique and then the participants will be asked to bring their leg to different positions. The test consists of five levels with each level increasing in difficulty.
Pelvic floor muscle function | change from baseline at 8 weeks
  Digital palpation will be used to evaluate pelvic floor muscle function while woman will be in the lithotomy position. Index + middle fingers will be inserted into the vagina.The women will be asked to squeeze these fingers in her vagina. force, endurance and speed parameters will be recorded.
Life Quality | change from baseline at 8 weeks
  King's Health Questionnaire will be used to evaluate life quality. It includes 9 sub-dimensions (General Health Perception, Incontinence Impact, Role Limitation, Physical Limitation, Social Limitation, Personal Limitation, Sleep/Energy Disturbance, Emotional Problems, and Severity Measures related UI). These sub-domains scores range from 0 to 100, where higher scores of indicate greater impairment in life quality
Perception of Recovery | after treatment (8th week)
  A 4-item Likert-type scale (worse, same, better, cured) will be used to evaluate perception of recovery
Compliance with recommendation | after treatment (8th week)
  Visual Analog Scale will be used to evaluate the compliance with recommendation.Participants were asked to rate compliance with recommendation on a 10 cm VAS line from 0 (not following recommendations at all) to 10 (completely following recommendations).

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Toprak Celenay, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Esenboğa Külliyesi, Turkey (Türkiye)